CLINICAL TRIAL: NCT01626794
Title: A Phase III Double Blind, Randomized, Multicenter, Controlled Study to Evaluate the Immunogenicity, Safety and Tolerability of VARIVAX Made With the Varicella Enhanced Process (VEP)
Brief Title: A Study to Evaluate the Immunogenicity, Safety, and Tolerability of VARIVAX™ Manufactured With a New Process (V210-062)
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: V210-062
Record Dates: First submitted 2012-06-08; First posted 2012-06-25 (Estimated); Last update posted 2015-01-27 (Estimated); Status verified 2015-01

CONDITIONS: Varicella
MeSH Terms: conditions — Chickenpox

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- VARIVAX™ VEP (Experimental)
  Interventions: Biological: VARIVAX™ VEP; Biological: M-M-R™ II
- VARIVAX™ 2007 Process (Active Comparator)
  Interventions: Biological: VARIVAX™ 2007 Process; Biological: M-M-R™ II

INTERVENTIONS:
Biological: VARIVAX™ VEP — Two 0.5 mL subcutaneous doses administered on Days 1 and 91
  Arms: VARIVAX™ VEP
Biological: VARIVAX™ 2007 Process — Two 0.5 mL subcutaneous doses administered on Days 1 and 91
  Arms: VARIVAX™ 2007 Process
Biological: M-M-R™ II — Two doses administered on Days 1 and 91 concomitantly with VARIVAX™ VEP or VARIVAX™ 2007 Process

SUMMARY:
This study will test the immunogenicity, safety, and tolerability of VARIVAX™ manufactured with the Varicella Enhanced Process (VEP) compared with the VARIVAX™ 2007 Process. The primary hypotheses being tested are 1)VARIVAX™ VEP will induce varicella-zoster virus (VZV) antibody responses that are non-inferior to those induced by VARIVAX™ 2007 process at 6 weeks after vaccination 1, and 2) VARIVAX™ VEP will induce an acceptable anti-VZV antibody response rate at 6 weeks after vaccination 1.

ELIGIBILITY:
Inclusion Criteria:

* negative clinical history of measles, mumps, rubella, varicella, and zoster

Exclusion Criteria:

* received any measles, mumps, rubella, or varicella vaccine at any time prior to the study, or is anticipated to receive any of these vaccines outside the study
* any congenital or acquired immune deficiency, neoplastic disease, or depressed immunity
* received systemic immunomodulatory steroids within 3 months prior to entering the study or is expected to require them throughout the study
* history of allergy or anaphylactoid reaction to neomycin, gelatin, sorbital, egg proteins, chicken proteins, or any components of M-M-R™ II or VARIVAX™
* received salicylates within 14 days prior to study vaccination
* exposed to measles, mumps, rubella, varicella, or zoster in the 4 weeks prior to study vaccination
* received any non-live vaccine within 14 days prior to any study vaccination or is expected to received such vaccine during the 42-day period after each study vaccination
* received any live vaccine within 30 days prior to any study vaccination or is expected to received such vaccine during the 42-day period after each study vaccination
* received immune globulin, a blood transfusion, or blood-derived products within 5 months prior to any study vaccination
* fever illness (≥102.2°F [39.0°C]) within 72 hours prior to study vaccination
* born to a human immunodeficiency virus (HIV)-infected mother
* participated in any other clinical trial (other than a surveillance study) within 30 days prior to study enrollment

Ages: 12 Months to 23 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2014-07; Primary Completion 2015-10 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Percent of Participants with VZV antibody levels ≥5 glycoprotein enzyme-linked immunosorbent assay (gpELISA) units/mL | Six weeks (43 days) after vaccination 1

SECONDARY OUTCOMES:
Percent of participants with fever (≥102.2°F [39.0°C] oral equivalent) | Days 1 to 42 after each vaccination
Percent of participants with measles-like, rubella-like, varicella-like, or zoster-like rash and mumps-like symptoms | Days 1 to 42 after each vaccination
Percent of participants with injection-site reactions | Days 1 to 5 after each vaccination